CLINICAL TRIAL: NCT02299258
Title: A Multicenter Randomized Controlled Trial of Malignant Gastric Outlet Obstruction: Tailored Partially Covered Stents (Placed Fluoroscopically) Versus Standard Uncovered Stents (Placed Endoscopically)
Brief Title: Gastric Outlet Obstructions Tailored Covered Stents for GOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Yuhang District (Other)
Responsible Party: Principal Investigator, Ding Shi, Dr., The First People's Hospital of Yuhang District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011ZHE008
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored stents MTN-WE-20/100-A (Active Comparator): The distal portion of the GOO tailored stents was semi-spherical, with a length of 20 mm, and a diameter of 28 mm. The middle segment had a diameter of 20 mm. The overall length of the stents was 100 mm. Both the middle part and the bottom of the proximal cup segment, and a part of the proximal funnel segment, were covered by a polyethylene membrane.
  Interventions: Device: Tailored stents MTN-WE-20/100-A
- Standard stents MTN-CG-s-20/100 (Experimental): Standard uncovered stents were used in the control group. The ends of the stents were semi-spherical with diameters of 28 mm and length of 20 mm. The length of the stents was 100 mm
  Interventions: Device: Standard stents MTN-CG-s-20/100

INTERVENTIONS:
Device: Standard stents MTN-CG-s-20/100 — The ends of the stents were semi-spherical with diameters of 28 mm and length of 20 mm. The length of the stents was 100 mm
  Arms: Standard stents MTN-CG-s-20/100
Device: Tailored stents MTN-WE-20/100-A — cup-shaped or funnel-shaped, according to the shapes of the proximal GOOs.
  Arms: Tailored stents MTN-WE-20/100-A

SUMMARY:
gastric outlet obstruction tailored versus standard stents for malignant gastric outlet obstruction treatments

DETAILED DESCRIPTION:
To determine the shape of the GOOs, stomach opacifications were performed using contrast media before stenting. In the GOO tailored group (33 cases), the distal stents were semi-spherical with a length of 20 mm and a diameter of 28 mm. The middle stent segments had diameters of 20 mm. The proximal ends of large cup-shaped stents had 53.3 ± 5.5 mm diameters and were 15 or 20 mm long, whereas the large funnel-shaped stents had 33.6 ± 3.6 mm diameters and were 25 or 30 mm long. The control group (32 cases) received standard uncovered stents (semi-spherical, with diameters of 28 mm and 20 mm long).Our hypothesis was that unresectable GOO tailored covered stents are superior to the standard uncovered ones in terms of stent re-obstruction and stent migration. In the current study the efficacy and safety of GOO tailored covered stents for the treatment of non-resectable GOOs caused by distal gastric cancer was compared with standard uncovered stents.

ELIGIBILITY:
Inclusion Criteria:

GOO defined by symptoms resulting in decreased oral intake (nausea, vomiting and inability to eat),the obstruction was caused by primary distal stomach cancer and the site of stenosis was between the gastric body and duodenum bulb

Exclusion Criteria:

the presence of only mild symptoms in patients who could tolerate a liquid diet, clinical evidence of perforation or peritonitis, evidence of multiple small-bowel obstructions because of peritoneal seeding as well as diabetes or other diseases that affect gastric motility and use of promotility agents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ding Shi, Study Director — The First People's Hospital of Yuhang District
Locations (1):
- The First People's Hospital of Yuhang District, Hangzhou, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tailored Stents MTN-WE-20/100-A | Standard Stents MTN-CG-s-20/100
Started | 32 | 31
Completed | 31 | 30
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Stents MTN-WE-20/100-A | Standard Stents MTN-CG-s-20/100 | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (7.7) | 75.8 (7.6) | 76.1 (7.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 32 | 31 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 18 | 16 | 34
Region of Enrollment [Number; unit: participants]
  China | 32 | 31 | 63
Gastric outlet obstruction score [Mean (Full Range); unit: units on a scale] — Gastric outlet obstruction score ranges from 2(best possible outcome) to 4(worst possible outcome)
  units on a scale | 3.2 [2.7 to 3.7] | 3.1 [2.7 to 3.5] | 3.2 [2.7 to 3.7]

OUTCOME MEASURES:

1. Primary Outcome: Efficiency of Stents
Description: number of participants considered having efficacious outcome. Efficacy is defined by Ingrowth + overgrowth in this study
Time Frame: up to 5 years
Measure: Number; unit: participants
Arm/Group | Tailored Stents MTN-WE-20/100-A | Standard Stents MTN-CG-s-20/100
Number analyzed (Participants) | 32 | 31
participants | 1 | 7

2. Secondary Outcome: Adverse Events
Description: bleeding, abdominal pain
Time Frame: up to 5 years
Measure: Number; unit: participants
Arm/Group | Tailored Stents MTN-WE-20/100-A | Standard Stents MTN-CG-s-20/100
Number analyzed (Participants) | 32 | 31
participants | 25 | 4

ADVERSE EVENTS:
Arm/Group | Tailored Stents MTN-WE-20/100-A | Standard Stents MTN-CG-s-20/100
Serious Adverse Events (participants affected / at risk) | 25/32 | 4/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored Stents MTN-WE-20/100-A (N=32) | Standard Stents MTN-CG-s-20/100 (N=31)
Bleeding (Blood and lymphatic system disorders) | 11 (11) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 1 (1)
Food impaction (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes